CLINICAL TRIAL: NCT03346265
Title: Progressive Modular Rebalancing (RMP) System Rehabilitation Combined With Sensory Cues for Rehabilitation of Patients With PD: a Randomized, Controlled Trial With Crossover.
Brief Title: Progressive Modular Rebalancing (RMP) System Rehabilitation Combined With Sensory Cues for Rehabilitation of Patients With PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Mariano Serrao, Clinical Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: s002
Record Dates: First submitted 2017-10-24; First posted 2017-11-17 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Parkinson Disease; Movement Disorders
Keywords: progressive modular rebalancing; PMR; visual sensory cues; SC; Parkinson Disease; Movement Disorders; Parkinson rehabilitation; neurocognitive method; motor performance; improving gait; physiotherapy; 3D motion analysis system; improvements
MeSH Terms: conditions — Parkinson Disease; Movement Disorders

STUDY DESIGN:
Intervention Model Description: Subjects participated in a baseline assessment session (T0, before rehabilitative treatment), followed by random allocation to 8 weeks of rehabilitative treatments (A or B) (T1), followed by 1 month of inactivity wash out period. Following this wash-out period, patients who received treatment A switched to the treatment B and viceversa. A computerized randomization schedule was generated on the computer and held by an investigator not involved in subject recruitment or assessment.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Treatment A consisted in a combined exercise program of 40 min duration RMP (Monari, 2004; Monari et al., 2016) and 20 min duration of gait training with sensory cues.
  RMP. RMP protocol was based on lengthening and muscular recruitment exercises by means of complex motor skills involving muscular kinetic chains in lower limbs and trunk. Each session was divided into muscular stretching exercise, aiming to increase step length and rotating trunk movements, and tailored progressive exercise therapy.
  Interventions: Other: Treatment A combined exercise program and gait training with sensory cues
- Group B (Experimental): Treatment B Conventional physiotherapy was composed of 4 sections of exercises, chiefly oriented to different body structures appropriate to movement (International Classification of Functioning, Disability and Health code): trunk (s760), pelvis (s750), lower extremity (s750), and upper extremity (s730) including shoulder region (s720). Domains focused on were (1) warm-up exercises, (2) trunk mobility exercises, (3) postural stability (b715), and (4) transferring oneself (d420) and changing body positions (d410).
  Interventions: Other: Treatment B Conventional physiotherapy

INTERVENTIONS:
Other: Treatment A combined exercise program and gait training with sensory cues — Treatment A consisted in a combined exercise program of 40 min duration RMP
  Arms: Group A
Other: Treatment B Conventional physiotherapy — Conventional physiotherapy was composed of 4 sections of exercises, chiefly oriented to different body structures appropriate to movement (International Classification of Functioning, Disability and Health code)
  Arms: Group B

SUMMARY:
In the present study, the investigators propose a rehabilitative program for Parkinson' disease based on the combination of a neurocognitive method, i.e. visual sensory cues, with a neurophysiological method, i.e. RMP, in a randomized controlled trial with cross-over. The rationale herein was that the RMP may globally improve patients in terms of trunk control, motor performance, muscle tone, endurance and so on, predisposing them to improvement of the gait rhythm and automaticity induced by use of the visual external cues.

The primary aim of this pilot, randomized, controlled, trial with crossover was to establish whether a 8-week exercise program focused at improving gait in people with PD was more effective than a same-duration program of standard physiotherapy. The secondary aim was to evaluate the effect on the disease's severity. At this aims investigators used a quantitative 3D motion analysis system to evaluate gait parameters and UPDRS-II and UPDR-III and H-Y staging to evaluate the severity of the disease.

The investigators hypothesised that the both exercise programs will improve standard physiotherapy, however the proposed program will yield better improvements for the people with PD.

DETAILED DESCRIPTION:
This study is a pilot, bi-centric, exploratory, randomized, controlled, crossover design with blind observer .

Subjects participated in a baseline assessment session (T0, before rehabilitative treatment), followed by random allocation to 8 weeks of rehabilitative treatments (A or B) (T1), followed by 1 month of inactivity wash out period. Following this wash-out period, patients who received treatment A switched to the treatment B and viceversa. A computerized randomization schedule was generated on the computer and held by an investigator not involved in subject recruitment or assessment.

Both clinical (neurological visit and scale administration) and instrumental (gait analysis) assessments were carried out 3 times: at baseline before rehabilitative treatment (T0), 4 weeks (T1, intermediate evaluation) and 8 weeks after rehabilitative treatments (T2, final evaluation). Medication was kept constant throughout the trial, and all interventions were performed at the same time of day for each patient during ON phase.

Participants were asked to maintain their pre-enrollment activity level and current medication dosage when not in the laboratory.

Assessors, for both clinical and instrumental evaluations, were blinded to the allocation treatment.

During the inactive condition, participants received usual care.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic PD according to UK bank criteria
* Hoehn and Yahr stages 1 to 3.
* United Parkinson Disease Rating Scale (UPDRS) gait subscore of 1 or more, no change in medication during the study period.
* All patients were in a stable drug program and had adapted to their current medications for at least 2 weeks.

Exclusion Criteria:

* cognitive deficits (defined as scores of <26 on the Mini-Mental State Examination [MMSE]),
* moderate or severe depression (defined as scores of >17 on the Beck Depression Inventory [BDI]),
* orthopedic and other gait-influencing diseases such as arthrosis or total hip joint replacement.

Ages: 55 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Stance phase duration ( change ) | - T0 baseline before rehabilitative treatment (T0) - T1 4 weeks (intermediate evaluation) - T2 8 weeks after rehabilitative treatments
swing phase duration ( change ) | - T0 baseline before rehabilitative treatment (T0) - T1 4 weeks (intermediate evaluation) - T2 8 weeks after rehabilitative treatments
double support phase duration ( change ) | - T0 baseline before rehabilitative treatment (T0) - T1 4 weeks (intermediate evaluation) - T2 8 weeks after rehabilitative treatments
cadence ( change ) | - T0 baseline before rehabilitative treatment (T0) - T1 4 weeks (intermediate evaluation) - T2 8 weeks after rehabilitative treatments
step length normalized for the leg length ( change ) | - T0 baseline before rehabilitative treatment (T0) - T1 4 weeks (intermediate evaluation) - T2 8 weeks after rehabilitative treatments
step length asymmetry ( change ) | - T0 baseline before rehabilitative treatment (T0) - T1 4 weeks (intermediate evaluation) - T2 8 weeks after rehabilitative treatments
step width ( change ) | - T0 baseline before rehabilitative treatment (T0) - T1 4 weeks (intermediate evaluation) - T2 8 weeks after rehabilitative treatments
mean speed ( change ) | - T0 baseline before rehabilitative treatment (T0) - T1 4 weeks (intermediate evaluation) - T2 8 weeks after rehabilitative treatments
maximal arm displacement on the posterior-anterior axis ( change ) | - T0 baseline before rehabilitative treatment (T0) - T1 4 weeks (intermediate evaluation) - T2 8 weeks after rehabilitative treatments
trunk Range of motion ( change ) | - T0 baseline before rehabilitative treatment (T0) - T1 4 weeks (intermediate evaluation) - T2 8 weeks after rehabilitative treatments

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | were carried out 3 times: at baseline before rehabilitative treatment (T0), 4 weeks (T1, intermediate evaluation) and 8 weeks after rehabilitative treatments (T2, final evaluation)
  * Part I: evaluation of mentation, behavior, and mood
  * Part II: self-evaluation of the activities of daily life (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food
  * Part III: clinician-scored monitored motor evaluation
  * Part IV: complications of therapy
Hoehn and Yahr | were carried out 3 times: at baseline before rehabilitative treatment (T0), 4 weeks (T1, intermediate evaluation) and 8 weeks after rehabilitative treatments (T2, final evaluation)
  1. Unilateral involvement only usually with minimal or no functional disability Unilateral involvement only 1.5 - Unilateral and axial involvement
  2. Bilateral or midline involvement without impairment of balance Bilateral involvement without impairment of balance 2.5 - Mild bilateral disease with recovery on pull test
  3. Bilateral disease: mild to moderate disability with impaired postural reflexes; physically independent Mild to moderate bilateral disease; some postural instability; physically independent
  4. Severely disabling disease; still able to walk or stand unassisted Severe disability; still able to walk or stand unassisted
  5. Confinement to bed or wheelchair unless aided Wheelchair bound or bedridden unless aided

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Serrao, PHD, Principal Investigator — Università "La Sapienza di Roma"
Locations (1):
- Policlinico Italia Srl, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keus SH, Munneke M, Nijkrake MJ, Kwakkel G, Bloem BR. Physical therapy in Parkinson's disease: evolution and future challenges. Mov Disord. 2009 Jan 15;24(1):1-14. doi: 10.1002/mds.22141. PMID 18946880
- [Background] Cassimatis C, Liu KP, Fahey P, Bissett M. The effectiveness of external sensory cues in improving functional performance in individuals with Parkinson's disease: a systematic review with meta-analysis. Int J Rehabil Res. 2016 Sep;39(3):211-8. doi: 10.1097/MRR.0000000000000171. PMID 27119224
- [Background] Westwater-Wood S, Adams N, Kerry R (2010): The use of proprioceptive neuromuscular facilitation in physiotherapy practice Physical Therapy Reviews Vol.15 No.1,p23-27
- [Background] Kabat H, Knapp ME (1943) The use of prostigmine in the treatment of poliomyelitis. JAMA 122: 989-995.
- [Background] Hove MJ, Keller PE. Impaired movement timing in neurological disorders: rehabilitation and treatment strategies. Ann N Y Acad Sci. 2015 Mar;1337(1):111-7. doi: 10.1111/nyas.12615. PMID 25773624
- [Background] Kisner, Carolyn & Colby, Lynn A. (2012):
- [Background] LEVINE MG, KABAT H. Proprioceptive facilitation of voluntary motion in man. J Nerv Ment Dis. 1953 Mar;117(3):199-211. doi: 10.1097/00005053-195303000-00002. No abstract available. PMID 13070034
- [Background] Monari G (2004) FNP, Facilitazioni Neurocinetiche Progressive. Elaborazione del concetto Kabat. Edi Ermes.
- [Background] Monari G (2013) RMP, Riequilibrio Modulare Progressivo. Elaborazione concetto Kabat. Edi Ermes
- [Background] Richards CL, Malouin F, Bedard PJ, Cioni M. Changes induced by L-DOPA and sensory cues on the gait of parkinsonian patients In: Woollacott M, Horak F, editors. Posture and gait: control mechanisms. XIth International Symposium of the Society for Postural and Gait Research, Portland, May 24-27, 1992. University of Oregon Books; 1992, p. 126-129.
- [Background] Marek SM, Cramer JT, Fincher AL, Massey LL, Dangelmaier SM, Purkayastha S, Fitz KA, Culbertson JY. Acute Effects of Static and Proprioceptive Neuromuscular Facilitation Stretching on Muscle Strength and Power Output. J Athl Train. 2005 Jun;40(2):94-103. PMID 15970955
- [Background] Sharman MJ, Cresswell AG, Riek S. Proprioceptive neuromuscular facilitation stretching : mechanisms and clinical implications. Sports Med. 2006;36(11):929-39. doi: 10.2165/00007256-200636110-00002. PMID 17052131
- [Background] McAtee RE, Charland J. Facilitated stretching: assisted and unassisted PNF stretching made easy. 2nd ed. Champaign (IL): Human Kinetics, 1999
- [Background] Kisner & Colby, p208,(2012)
- [Background] Kisner & Colby 2012, p208
- [Background] Nagarwal, A.K., Zutshi K., Ram C.S., Zafar R.(2010). Improvement of hamstring flexibility: A comparison between two PNFstretching techniques. International Journal of Sports Science and Engineering.4 (2010) 1, pp 025-033
- [Background] Surburg PR, Schrader JW. Proprioceptive neuromuscular facilitation techniques in sports medicine: a reassessment. J Athl Train. 1997 Jan;32(1):34-9. PMID 16558430
- [Background] Feland JB, Marin HN. Effect of submaximal contraction intensity in contract-relax proprioceptive neuromuscular facilitation stretching. Br J Sports Med. 2004 Aug;38(4):E18. doi: 10.1136/bjsm.2003.010967. PMID 15273211
- [Background] Ford P, McChesney J. Duration of maintained hamstring ROM following termination of three stretching protocols. J Sport Rehabil. 2007 Feb;16(1):18-27. doi: 10.1123/jsr.16.1.18. PMID 17699884
- [Background] Nagarwal, A.K., Zutshi K., Ram C.S., Zafar R. (2010). Improvement of hamstring flexibility: A comparison between two PNF stretching techniques. International Journal of Sports Science and Engineering. 4 (2010) 1, pp 025-033.
- [Background] Kavanagh J, Barrett R, Morrison S. The role of the neck and trunk in facilitating head stability during walking. Exp Brain Res. 2006 Jul;172(4):454-63. doi: 10.1007/s00221-006-0353-6. Epub 2006 Feb 18. PMID 16489437
- [Derived] Serrao M, Pierelli F, Sinibaldi E, Chini G, Castiglia SF, Priori M, Gimma D, Sellitto G, Ranavolo A, Conte C, Bartolo M, Monari G. Progressive Modular Rebalancing System and Visual Cueing for Gait Rehabilitation in Parkinson's Disease: A Pilot, Randomized, Controlled Trial With Crossover. Front Neurol. 2019 Aug 29;10:902. doi: 10.3389/fneur.2019.00902. eCollection 2019. PMID 31543859